CLINICAL TRIAL: NCT03179969
Title: Interventional Therapy of Paravalvular Post-surgical or Post-interventional Valve Replacement Leaks With Plug Devices: The German Plug - Registry
Brief Title: The German Plug - Registry
Acronym: PLUG
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: PLUG Registry
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-05

CONDITIONS: Heart Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: paravalvular leak — Observational study on patients with paravalvular leak

SUMMARY:
In approximately 10-15% of all patients after surgical or interventional heart valve replacement, flapping defects appear as complications in the long-term course, so-called paravalvular / paraprothetic leaks (PVL). In some patients, due to the severity of the defect, a new procedure is required - with a not inconsiderable disease or even mortality risk

DETAILED DESCRIPTION:
In approximately 10-15% of all patients after surgical or interventional heart valve replacement, flapping defects appear as complications in the long-term course, so-called paravalvular / paraprothetic leaks (PVL). In some patients, due to the severity of the defect, a new procedure is required - with a not inconsiderable disease or even mortality risk. For a number of years, the catheter-based closure of the defect has been increasingly used by means of the implantation of plug-devices as a new treatment method for patients with a high surgical risk. The existing data on the operation method and safety of the method already used at some centers are promising. In order to demonstrate the clinical routine of patients with an interventional occlusion of a PVL in a timely manner, the Stiftung IHF Ludwigshafen will publish a multicentric register entitled "Deutsches Plug Register" The goal is, among other things, the documentation of patient characteristics, indications, and complications of treated patients.The German Heart Foundation promotes the setting up of the plug register.

In this time, 200 patients with valve prosthesis defects, with which the indication for plug implantation was placed prospectively and retrospectively, are to be included in the register.

ELIGIBILITY:
Inclusion Criteria:

* heart valve replacement
* Valve Replacement Leaks
* Plug Device

Exclusion Criteria:

* no written consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 200 patients with valve prosthesis defects, with which the indication for plug implantation was placed prospectively and retrospectively, are to be included in the register.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
mortality risk | five years
  observation of the mortality risk

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Zahn, Prof., Study Chair — Klinikum Ludwigshafen
Locations (1):
- Klinikum Ludwigshafen, Ludwigshafen, Deutschland, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Konrad H, Werner N, Ouarrak T, Schofer J, Lubos E, Geist V, Eggebrecht H, Butter C, Schmitz T, Schafer U, Schumacher B, Schneider S, Zeymer U, Zahn R. Acute and long-term results of interventional treatment of paravalvular leaks after prosthetic valve replacement with plug devices: results from a prospective multicentre registry. Clin Res Cardiol. 2025 Jun 2. doi: 10.1007/s00392-025-02681-w. Online ahead of print. PMID 40455223